CLINICAL TRIAL: NCT02851394
Title: Evaluation Of The Efficacy Of A Bolus Infiltration Of The Anaesthetic Tramadol Associated With Continuous Local Anaesthesia Administered Via A Wound Catheter Following Heart Surgery Via Sternotomy At Dijon Chu Single-Centre, Double-Blind, Randomized, Controlled Clinical Trial
Brief Title: Advantage of Tramadol in Local Analgesia Post-Sternotomy
Acronym: ATLAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bethenod Ellouze 2014
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Heart Surgery Via Sternotomy; Post-operative Analgesia
MeSH Terms: interventions — Levobupivacaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Levobupivacaine group (Active Comparator)
  Interventions: Drug: Levobupivacaine
- Levobupivacaine + tramadol group (Experimental)
  Interventions: Drug: levobupivacaine; Drug: tramadol

INTERVENTIONS:
Drug: Levobupivacaine
  Arms: Levobupivacaine group
Drug: levobupivacaine
  Arms: Levobupivacaine + tramadol group
Drug: tramadol
  Arms: Levobupivacaine + tramadol group

SUMMARY:
Sternotomy, the reference approach for heart surgery, may induce profound and intense post-operative pain. One method of analgesia used is patient-controlled intravenous morphine.

The analgesic efficacy of continuous wound infiltration at the sternum following heart surgery has been demonstrated.

The analgesic catheter placed near the sternotomy wound reduces the consumption of morphine.

The aim of this study is to determine whether a bolus of tramadol associated with the continuous administration of levobupivacaine via the wound catheter could potentiate the local anaesthetic effects, thus leading to a decreased consumption of postoperative intravenous morphine, and a decrease in morphine-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written consent
* Patients over 18 years old
* Patients undergoing heart surgery via sternotomy: aortic valve surgery, mitral valve surgery, tricuspid valve surgery, atrial myxoma, coronary artery bypass graft, aorta surgery
* Patients undergoing emergency or scheduled surgery

Exclusion Criteria:

* Adults under guardianship
* Persons without national health insurance cover
* Pregnant or breast-feeding women
* Patients already included in the study once
* Patients with aortic dissection
* Patients with mediastinitis or sternal nonunion
* Patients undergoing heart surgery for the second or more time
* Patients with local infection or generalized bacteraemia-type infection
* Patients with hypersensitivity to local anaesthetics or to tramadol or to opiates or to one of the excipients present in the products used
* Patients with hypersensitivity to paracetamol or to paracetamol hydrochloride (prodrug of paracetamol)
* Patients on antidepressants, gabapentin, pregabalin, neuroleptics
* Patients with a history of convulsions or epilepsy
* Patients with preoperative cognitive dysfunction
* Patients with intracranial hypertension
* Chronic use of morphines or high-dose steroid or non-steroid anti-inflammatory agents
* Patients with acute or chronic kidney failure (creatininemia > 170 µmol/L)
* Patients with liver failure or porphyria
* Patients under 17 years old
* Patients with severe respiratory failure
* Patients treated with a non-selective MAOI (iproniazid), a selective MAOI A (moclobemid, toloxatone), selective MAO-B inhibitor (Selegiline) or linezolid (Zyvoxid®)
* Patients with acute intoxication or an overdose of products that depress the central nervous system (alcohol, hypnotics, other analgesics…)
* Patients with severe hypotension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Consumption of morphine, expressed in milligrams, in the post-operative period | 48 hour after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Bethenod F, Ellouze O, Berthoud V, Missaoui A, Cransac A, Aho S, Bouchot O, Girard C, Guinot PG, Bouhemad B. A single dose of tramadol in continuous wound analgesia with levobupivacaine does not reduce post-sternotomy pain: a randomized controlled trial. J Pain Res. 2019 Sep 18;12:2733-2741. doi: 10.2147/JPR.S211042. eCollection 2019. PMID 31571977